CLINICAL TRIAL: NCT04357678
Title: Comparison of Qui Gong Programme With Short Form Sun Style Tai Chi in COPD Patients
Brief Title: Qui Gong Programme vs Short Form Sun Style Tai Chi in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00590 Qurrat ul Ain
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: COPD
Keywords: Pulmonary Disease; Qigong; Tai chi
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qi Gong Programme (Experimental): Qi Gong Programme
  Interventions: Other: Qi Gong Programme
- Short Form Sun Style Tai Chi (Experimental): Short Form Sun Style Tai Chi
  Interventions: Other: Short Form Sun Style Tai Chi

INTERVENTIONS:
Other: Qi Gong Programme — Warm-up: In warm up session joint activities were performed along with light stretching. Patients performed these activities with instructor's commands for 5 minutes.
  Liu Zi Jue exercise: patients performed intact Liu Zi Jue exercise (form of Qigong).
  This includes six healing sounds, Xu, He, Hu, Si, Chui, Xi and the Harmonized actions along with the instructor for 20 minutes. Cooling-down: After completion of Qigong, patient done gentle stretching to adjust back their breathing and this cool down session lasted for 5 minutes. Subjects received supervised training session for 30 min twice a week.
  Arms: Qi Gong Programme
Other: Short Form Sun Style Tai Chi — Commencing Movement, Opening and closing hand, Single whip, Waving hands in the cloud, Opening and closing hands, Brush knee, Playing lute, Perry and Punch, Block and close, Pushing the mountain, Closing movement.
  Participants attended two supervised 30min sessions twice a week. Participants learnt 3 to 4 forms per week and at the completion of study (which is the six week of training), they completed all 21 forms. In each training session, participants revised previous SSTC forms that they learnt earlier up to that session.
  Arms: Short Form Sun Style Tai Chi

SUMMARY:
This was a Randomized control Trial. Purposive sampling was done to obtained Sample (n=78) which were randomly allocated to Group A (n=39) and Group B (n=39). Study was conducted from August 2019 to December 2019 in HBS Hospital Islamabad.To determine the effects of Qigong vs. Shot form Sun Style Tai Chi (SSTC) on Lung function, six min walk distance, dyspnea and quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by persistent respiratory symptoms and air-ﬂow limitation. Dyspnea is related with daily life activity. COPD patients often suffer from dyspnea and exacerbation, which leads to inactivity, deconditioning, and poor functional capacity and quality of life. Several interventions have been investigated with the aim of improving lung function, decreasing dyspnea symptoms and improving quality of life in this patient.

Tai Chi, an exercise involving both upper and lower extremities, originated from China. Tai chi is characterized by posture alignment, weight shifting and circular movements that incorporate elements of muscle endurance and strengthening, balance, relaxation and breathing control. Among previous studies Tai Chi in pulmonary rehabilitation showed a modest complementary benefit in exercise capacity.

The Tai Chi program is a safe, effective and feasible method to improve exercise capacity and health-related quality of life in people with COPD. Short form sun style Tai chi is one of the most common styles of t'ai chi. each form can be broken down into several movements which make it easy to learn and teach. Compared to some other styles of t'ai chi, SSTC involves less difficult movements, such as less deep-knee bending and single leg standing, which may make it more suitable for older people.

Qi Gong is defined as a mind-body exercise that involves whole body movements, breathing techniques, postural control, and internal awareness.

effects of Qi Gong on functional capacity and lung functions in COPD patients , and concluded that functional capacity, dyspnea scores and quality of life was significantly improved in mild to moderate COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Diagnosed patient: Mild to moderate stage COPD according to GOLD criteria {i-e Global Initiative for Chronic Obstructive Lung Disease (GOLD) }
* Patients who can walk without any dependency were included in study.

Exclusion Criteria:

* Patients with acute exacerbation within 4 weeks before starting the study
* Patient having significant, cognitive impairment
* Patient having Tuberculosis, asthma
* Patient having musculoskeletal
* Patient having psychological, cardiovascular and benign conditions (that prohibit exercise were excluded from the study)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6th week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
6 min walk test: Distance (meters) | 6th week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale (mMRC) | 6 week
  Changes from the Baseline, It was used to measure Dyspnea score. This scale ranges from 0 to 4 in which 0 indicates that strenuous exercise leads to breathlessness" and 4 means "too breathless"
Quality of life: St. George's Respiratory Questionnaire (SGRQ) | 6 week
  was used to access the quality of life; SGRQ is used for determining quality of life in COPD patients. This questionnaire is designed in 50 items to check the impact of COPD. 0 to 100 is the range of this score. Scores having higher values means more limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- HBS General Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Lee A, Lee DT, Suen LK, Tam WW, Chair SY, Griffiths P. The sustaining effects of Tai chi Qigong on physiological health for COPD patients: a randomized controlled trial. Complement Ther Med. 2013 Dec;21(6):585-94. doi: 10.1016/j.ctim.2013.09.008. Epub 2013 Oct 8. PMID 24280465
- [Background] Chan AW, Lee A, Suen LK, Tam WW. Effectiveness of a Tai chi Qigong program in promoting health-related quality of life and perceived social support in chronic obstructive pulmonary disease clients. Qual Life Res. 2010 Jun;19(5):653-64. doi: 10.1007/s11136-010-9632-6. Epub 2010 Mar 15. PMID 20229333
- [Background] Wu LL, Lin ZK, Weng HD, Qi QF, Lu J, Liu KX. Effectiveness of meditative movement on COPD: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 Apr 17;13:1239-1250. doi: 10.2147/COPD.S159042. eCollection 2018. PMID 29713157
- [Background] Zhu S, Shi K, Yan J, He Z, Wang Y, Yi Q, Huang H. A modified 6-form Tai Chi for patients with COPD. Complement Ther Med. 2018 Aug;39:36-42. doi: 10.1016/j.ctim.2018.05.007. Epub 2018 May 17. PMID 30012390
- [Background] Lorna Ng LK, Raymond Tang ,Cheetham Siu, Lawrence Fung, Albert Lee, Wilson Tamd. Effectiveness of incorporating Tai Chi in a pulmonary rehabilitation program for Chronic Obstructive Pulmonary Disease (COPD) in primary care-A pilot randomized controlled trial. European Journal of Integrative Medicine2015;6(3): 248-58.
- [Background] Nagaratnam N. NK, Cheuk G. Chronic Obstructive Pulmonary Disease (COPD). Geriatric Diseases 2018
- [Background] Leung RW, McKeough ZJ, Peters MJ, Alison JA. Short-form Sun-style t'ai chi as an exercise training modality in people with COPD. Eur Respir J. 2013 May;41(5):1051-7. doi: 10.1183/09031936.00036912. Epub 2012 Aug 9. PMID 22878879
- [Background] Regina Wai Man Leung*, Zoe J. McKeough, Matthew J. Peters
- [Background] Kantatong T, Panpanich R, Deesomchok A, Sungkarat S, Siviroj P. Effects of the tai chi qigong programme on functional capacity, and lung function in chronic obstructive pulmonary disease patients: A ramdomised controlled trial. J Tradit Complement Med. 2019 Apr 1;10(4):354-359. doi: 10.1016/j.jtcme.2019.03.008. eCollection 2020 Jul. PMID 32695652
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278